CLINICAL TRIAL: NCT06835634
Title: PANDA, Progressive Advancements in Neurosurgery, Data and Analysis Database
Brief Title: Progressive Advancements in Neurosurgery, Data and Analysis Database
Acronym: PANDA
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7202
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Spine Disease; Central Nervous System Diseases; Peripheral Nervous System Diseases
MeSH Terms: conditions — Spinal Diseases; Central Nervous System Diseases; Peripheral Nervous System Diseases | interventions — Psychological Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Self reported questionnaires — PROMs and psychological tests submission in patients affected by neurosurgical diseases
  Other Names: psychological tests

SUMMARY:
Neurosurgical diseases encompass a highly heterogeneous group of conditions, including oncological, malformative, traumatic, spinal, vascular, infectious diseases, and cerebrospinal fluid dynamics disorders. Several systematic reviews on the level of evidence in neurosurgical diseases have documented the low percentage of high-quality scientific evidence in this field of medicine. Clinical practice is strongly influenced by individual physician preferences, leading to significant heterogeneity among different centers both in Italy and internationally. This overall picture highlights the need for tools that can accurately characterize the numerous diagnostic variables influencing therapeutic outcomes in patients with neurosurgical diseases.

Primary Objective To establish a prospective data collection of adult patients with neurosurgical diseases, providing real-life data on the current management of patients at the Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome and the participating centers.

Secondary Objectives To create a database of adult patients with neurosurgical diseases who may be potential candidates for enrollment in clinical trials.

To conduct observational research on neurosurgical diseases, particularly in cases where no curative treatment options are currently available.

To identify potential predictors of poor outcomes or treatment response. To assess the clinical history and treatment response of patients, including for internal audit purposes (e.g., supporting Morbidity & Mortality conferences).

To provide support for the development and monitoring of quality indicators related to patient care.

ELIGIBILITY:
Inclusion Criteria:

* Age at first contact equal to or greater than 18 years at the time of informed consent signature.
* Diagnosis of a neurosurgical disease.

Exclusion Criteria:

* Refusal to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population affected by a **neurosurgical disease** at the time of **first contact with the patient**, whether in an **outpatient or inpatient setting**, at the facilities of the centers participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 7500 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2035-02-10 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Data collection of adult patients with neurosurgical diseases | 1 year
  To establish a prospective data collection of adult patients with neurosurgical diseases, providing real-life data on the current management of patients at the Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome and the participating centers.

SECONDARY OUTCOMES:
database of adult patients with neurosurgical diseases | 1 year
  To create a database of adult patients with neurosurgical diseases who may be potential candidates for enrollment in clinical trials.
observational research on neurosurgical diseases | 1 year
  To conduct observational research on neurosurgical diseases, particularly in cases where no curative treatment options are currently available.
potential predictors of treatment response | 1 year
  To identify potential predictors of poor outcomes or treatment response
development and monitoring of quality indicators | 1 year
  To provide support for the development and monitoring of quality indicators related to patient care.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Olivi, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, UOC Neurochirurgia, Roma, Italy